CLINICAL TRIAL: NCT01842412
Title: The Initial Effect of Training on Mitochondrial Function in Patients With Intermittent Claudication
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/395/REK midt
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Intermittent Claudication
Keywords: Mitochondria, Muscle; Exercise
MeSH Terms: conditions — Intermittent Claudication; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- claudication
  Interventions: Behavioral: exercise
- healthy
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — one bout of exercise training

SUMMARY:
The hypothesis of this study is that one bout of leg exercise gives acute qualitative changes in mitochondrial function in claudication. Final purpose is to determine the optimal exercise frequency in treatment of claudication.

ELIGIBILITY:
Inclusion Criteria:

* A history of any type of uni- or bilateral exertion leg pain.
* A maximal claudication distance that is less than 300 meter
* Diagnosed with intermittent claudication secondary to vascular insufficiency
* An ankle-brachial index between 0.4 and 0.9.
* Lives in Trondheim

Exclusion Criteria:

* Diagnosed with critical limb ischemia
* ankle-brachial index > 0.90 or < 0.4
* Limited exercise tolerance
* Warfarin or heparin usage
* Diabetes mellitus
* Underwent a vascular intervention in the last 3 months
* Active cancer, renal- or liver disease.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic, vascular surgery, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function | One day
  respirometry

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ellingsen, prof, Study Director — Norwegisn University of Science and Technology
Locations (1):
- Department for circulation and medical imaging, NTNU, Trondheim, Postboks 8905, Norway

REFERENCES:
- [Result] van Schaardenburgh M, Wohlwend M, Rognmo O, Mattsson EJ. Mitochondrial Respiration after One Session of Calf Raise Exercise in Patients with Peripheral Vascular Disease and Healthy Older Adults. PLoS One. 2016 Oct 19;11(10):e0165038. doi: 10.1371/journal.pone.0165038. eCollection 2016. PMID 27760222